CLINICAL TRIAL: NCT00169117
Title: A Stitch in Time May Save Lives: Turning Poor Bednets Into Good Ones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Durham (Other); Medical Research Council Unit, The Gambia (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DIF8
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
Keywords: Mosquito nets; Malaria prevention; Songs; Posters; Net repair; Bednets
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Behavioural intervention: Songs/posters aimed at behaviour change to increase repair and maintenance of mosquito nets
  Interventions: Behavioral: Songs/posters aimed at behaviour change

INTERVENTIONS:
Behavioral: Songs/posters aimed at behaviour change — This was a behavioural intervention, using songs and posters composed/designed by community members which aimed at behaviour change to increase repair and maintenance of mosquito nets

SUMMARY:
Although the use of mosquito nets has increased in Africa, many of the nets used are in a poor state, and not an effective barrier against mosquitoes. This pilot study examines whether subsistence farmers in rural Africa can be encouraged to repair their mosquito nets and use their bednets appropriately. Attitudes and practises on sewing and net use were examined in The Gambia and an intervention developed to promote net repair. Songs and posters were used to emphasise the importance of repairing nets and their correct use, and served as aural and visual reminders to repair nets now rather than postpone this household chore. The intervention was aimed at effectively and cheaply turning a poor net into a good one.

DETAILED DESCRIPTION:
Sleeping under an insecticide-treated net protects the sleeper from mosquito bites and is highly effective means of reducing the risk of malaria. Recent studies in The Gambia and Kenya have shown that untreated bednets in good condition can also protect against malaria (51% protection against parasitaemia, 95% CIs 34-64%). However, most children in rural Gambia sleep under untreated nets in poor condition, often with a few holes, and do not close their nets properly at night. These children remain exposed to mosquito bites and the risk of malaria.

This pilot study examines whether subsistence farmers in rural Africa can be encouraged to repair their mosquito nets and use their bednets appropriately. Attitudes and practises on sewing and net use were examined in rural Gambia and an intervention developed to promote net repair. Songs and posters were used to emphasise the importance of repairing nets and their correct use, and served as aural and visual reminders to repair nets now rather than postpone this household chore. The intervention was aimed at effectively and cheaply turning a poor net into a good one.

The intervention was developed and implemented in two neighbouring villages in The Gambia, with each village composing their own songs. There was no formal control village. An internal comparison group was used in which the nets of responders and non-responders living within the same village were compared.The success of the intervention was assessed by: recording the number of nets repaired and used correctly for malarial prevention before and after the intervention; by counts of mosquitoes entering the nets classified according to number of holes and degree of repair; as well as by canvassing participants' opinions.

ELIGIBILITY:
Inclusion Criteria:

* Community consent
* Willingness to participate in study

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 772 (Actual)
Dates: Start 2002-06; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Number of bednets repaired (pre- vs post intervention) | November 2003
Mean proportion of holes repaired/net (pre- vs post intervention) | November 2003
Reduction in mosquitoes with a good net compared with a poor one (pre-intervention survey). | November 2003
Reduction in mosquitoes with a good net compared with a repaired net (post-intervention survey) | November 2003

SECONDARY OUTCOMES:
Community acceptability | November 2003

CONTACTS AND LOCATIONS:
Overall Officials: Steven W Lindsay, PhD, Principal Investigator — University of Durham; Sian E Clarke, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine, University of London, UK; Catherine Panter-Brick, PhD, Principal Investigator — University of Durham
Locations (1):
- Medical Research Council Laboratories, Farafenni, The Gambia

REFERENCES:
- [Background] Lomas H, Panter-Brick C, Clarke S, Lindsay S, Pinder M & Walraven G. (2004). A community intervention to repair bed nets for malaria prevention in the Gambia [abstract]. Annals of Human Biology, 31(1): 116
- [Result] Panter-Brick C, Clarke SE, Lomas H, Pinder M, Lindsay SW. Culturally compelling strategies for behaviour change: a social ecology model and case study in malaria prevention. Soc Sci Med. 2006 Jun;62(11):2810-25. doi: 10.1016/j.socscimed.2005.10.009. Epub 2005 Dec 13. PMID 16352385